CLINICAL TRIAL: NCT00051740
Title: Compensating for Cognitive Deficits in Schizophrenia
Brief Title: Treating Thought Problems in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dawn Velligan, Clinical Professor Department of Psychiatry, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH061775 (NIH); DATR A4-GPS
Record Dates: First submitted 2003-01-15; First posted 2003-01-17 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cognitive Adaptation Therapy (Active Comparator): Subjects receive Cognitive adaptation therapy as part of treatment for schizophrenia
  Interventions: Behavioral: Cognitive Adaptation Therapy (CAT)
- Minimal Environmental Support (Active Comparator): Subjects receive minimal environmental support in schizophrenia treatment
  Interventions: Behavioral: Minimal Environmental Supports (MES)

INTERVENTIONS:
Behavioral: Cognitive Adaptation Therapy (CAT)
  Arms: Cognitive Adaptation Therapy
Behavioral: Minimal Environmental Supports (MES)
  Arms: Minimal Environmental Support

SUMMARY:
This study will compare Cognitive Adaptation Training (CAT) to minimal schizophrenia treatment. This study will also determine whether the intensity of CAT can be reduced and still provide benefits to patients with schizophrenia.

DETAILED DESCRIPTION:
Many schizophrenia patients have serious difficulties that affect their quality of life. Cognitive Adaptation Training (CAT) may improve adaptive functioning, quality of life, and rates of relapse in schizophrenia patients. CAT, which involves compensatory strategies or environmental supports, is tailored to each individual and is based on executive functioning levels and other factors.

Participants are randomly assigned to CAT, Minimal Environmental Supports (MES), or treatment as usual for 2 years. Participants receiving CAT will have a trained therapist make weekly visits to their home for 9 months. Over the following 3 months, the frequency of CAT visits will be slowly reduced to once a month. For the remaining 12 months of treatment, patients receive CAT only once a month.

Participants assigned to the MES group receive a generic set of supplies and equipment (calendar, alarm clock, watch, bus passes, etc.) at the beginning of the 2-year period. Each month, the supplies are replenished as necessary during the patient's scheduled clinic visit.

In all groups, assessments of adaptive function and quality of life occur at study start and at 3, 6, 9, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Treatment with an atypical antipsychotic medication
* Stable living environment
* Able to read, understand, and complete rating scales and neuropsychological testing
* Willing to participate in psychosocial treatments for schizophrenia that may involve home visits

Exclusion Criteria:

* History of significant head trauma, seizure disorder, or mental retardation
* Alcohol or drug abuse that could interfere with participation in the study
* Treatment by an ACT team
* History of violence in the past year
* Score > 80 on the SOFAS
* Hospitalized in the past year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Primary | up to 24 months
  compare Cognitive Adaptation Training (CAT) to minimal schizophrenia treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I. Velligan, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States